CLINICAL TRIAL: NCT04259216
Title: Intervention Media to Prevent Adolescent Cyber-conflict Through Technology
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0000000136/132580194; 0000000136/132580194 (Other Grant/Funding Number: University of Wisconsin Madison/PIVOTAL)
Record Dates: First submitted 2020-01-30; First posted 2020-02-06 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2020-12

CONDITIONS: Cyberbullying
Keywords: cyber-victimization; mobile application; mhealth; remote intervention
MeSH Terms: conditions — Cyberbullying

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPACT Intervention (Experimental): 1. Remote brief video session, introducing basic principles of cognitive behavioral theory and the structure of the mobile application message portion of the intervention.
  2. Eight-weeks longitudinal tailored Cognitive Behavioral Therapy (CBT)-based messaging program
  Interventions: Behavioral: IMPACT Intervention
- Control Enhanced Online Resources (EOR) (Active Comparator): 1. We will provide a link to an online resource packet with information on bullying and mental health resources.
  Interventions: Other: Control: Enhanced Online Resources (EOR)

INTERVENTIONS:
Behavioral: IMPACT Intervention — Brief remote session + tailored, daily 8-week mobile application facilitated messaging secondary prevention intervention.
  Arms: IMPACT Intervention
Other: Control: Enhanced Online Resources (EOR) — EOR group participants will receive standardized information on cyberbullying.
  Arms: Control Enhanced Online Resources (EOR)

SUMMARY:
The purpose of this randomized pilot trial is to test the feasibility of online recruitment and intervention delivery of the same Intervention to Prevent Cyber-victimization among Adolescents through Text-Messaging (iPACT) intervention content, delivered via mobile app (instead of SMS). This study includes a brief remote introductory session, followed by eight weeks of daily, tailored two-way messages, with an 8-week assessment. If successful, the IMPACT intervention will demonstrate feasibility and acceptability of an easily disseminable intervention to improve wellness and resilience among at-risk youth and their social network.

DETAILED DESCRIPTION:
Cyber-bullying, defined as intentional harm of others through computers, cellphones, and other electronic devices, is increasingly common. Approximately one quarter of American adolescents report that they have been cyber-victims in the past year (with rates ranging from 6-72%, depending on the study). Being a victim of cyber-bullying is strongly associated with multiple negative consequences. Cyber-victimization predicts depressive symptoms and suicidality; it correlates with Post Traumatic Stress Disorder (PTSD) symptoms, alcohol and other drug use, physical peer violence, and dating violence. Emotional regulation skills and positive social supports may be protective. Development of an acceptable, effective, and potentially disseminable secondary prevention tool, to decrease both the frequency and consequences of cyber-victimization, is therefore of high public health importance.

Effective, acceptable, and easily disseminable secondary prevention tools are needed to improve adolescent resilience and reduce the negative effects of cybervictimization. Ninety-five percent of adolescents have access to a smartphone. Our team recently conducted an NICHD-funded pilot of an in-person brief intervention + automated 8-week interactive text-message program ("iPACT"), to reduce cyber-victimization among youth recruited in a pediatric clinic. Pilot testing of iPACT showed high acceptability (89% responses to daily messages), and preliminary signals of efficacy (e.g. improved use of bystander behaviors). However, our team identified two elements for improvement. First, the in-person brief intervention was difficult to deliver during a clinic visit due to patients' time limitations. Second, our and others' work suggests that at-risk youth are more commonly witnesses of cyber-victimization, than victims themselves, and therefore need greater content focused on bystander intervention. Third, at-risk youth may be more easily identified online than in person.

Participants will be identified through targeted Instagram advertisements. If eligible, participants will complete an online assent form followed by a series of comprehensive questions to assess for capacity to assent. Participants will complete a baseline assessment and will be randomized to experimental (IMPACT, n=40) or connection to Enhance Online Resources (EOR, n=40).

This study will pilot an enhanced intervention, "IMPACT" is a two-part remotely-delivered intervention for youth reporting online victimization, derived from iPACT's existing structure, to promote pro-social behavior and enhance wellness among at-risk adolescents. We will deliver a brief, computer-guided discussion (an adaptation of iPACT's in-person intervention) remotely via video chat; and deliver 8 weeks of automated, enhanced message content that helps participants identify, intervene in, and effectively reduce the impact of witnessed or experienced cyberbullying. EOR group participants will receive standardized information on cyberbullying.

Participants will complete assessments at baseline, 8 weeks, and 16 week to measure cyberbullying, peer violence, and cognitive/behavioral skill sets. At the 8 week follow-up, we will assess for efficacy, acceptability, usability, and feasibility through standardized qualitative and quantitative measures.

ELIGIBILITY:
Inclusion Criteria:

* reside in the US
* being English-speaking
* having a English-speaking parent
* active Instagram account
* self-reporting cyber-victimization (defined as endorsing >1 past-year episode of technology mediated victimization)

Exclusion Criteria:

* being cognitively unable to take part in the intervention as determined by study staff

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-05-03 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability: Enrollment Rate | Baseline
  % of eligible participants who consented and completed enrollment
Intervention Acceptability: Participant Satisfaction | 8 week post-enrollment
  % of participants that agree or strongly agree on the quantitative acceptability assessment and qualitative interviews
Intervention Feasibility: Participant Engagement | Baseline to 8 weeks post-enrollment (close of intervention)
  % of intervention participants that complete study components including responding to at least one of the daily message queries, and how many requested on-demand support messages

SECONDARY OUTCOMES:
Cyber-victimization and related online behaviors | Baseline, 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment
  Change in University of New Hampshire Internet Safety Education Survey (UNH) from enrollment other forms (cyberbullying); investigators selected 5 items from the survey to measure. Items are scored by participants' self-report of online harassment experiences ranging from 0 ("Never") to 4 ("7 or more times"). Possible score range of 0-20, with higher scores indicating greater number of online harassment experiences.
Psychological stress | Baseline, 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment
  Change in Patient-Reported Outcomes Measurement Information System (PROMIS); Four items are scored by participants' self-report of Psychological Stress ranging from 1 ("Never") to 5 ("Always"). The raw score ranges from 4 to 20, 4 representing least and 20 representing most psychological stress.
Positive affect | Baseline, 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment
  Change in Patient-Reported Outcomes Measurement Information System (PROMIS); Four items are scored by participants' self-report of Positive Affect ranging from 1 ("Never") to 5 ("Always"). The raw score ranges from 4 to 20, 4 representing least and 20 representing most positive affect.
Well-being Index | Baseline, 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment
  The World Health Organization- Five- Well-Being Index (WHO-5 ) from enrollment other forms (well-being); Five items are scored by participants' self-report of well-being ranging from 0 ("At no time") to 5 ("All of the time"). The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.
Theoretical mechanisms of prosocial behaviors and self-efficacy | Baseline, 8 weeks post-enrollment (close of intervention), 16 weeks post-enrollment
  Change in Bystander Intervention in Bullying Measures; 5 items from the Bystander Intervention in Bullying Measures and 8 items from the University of New Hampshire Internet Safety Education Survey. Items are scored by participants' self-report of online bystander behavior ranging from 1 ("Strongly disagree") to 5 ("Strongly agree"). Possible score range of 13-65, with higher scores indicating greater personal responsibility/self-efficacy to intervene when witnessing online harassment experiences (prosocial behavior and self-efficacy).

CONTACTS AND LOCATIONS:
Overall Officials: Megan Ranney, MD MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kutok ER, Dunsiger S, Patena JV, Nugent NR, Riese A, Rosen RK, Ranney ML. A Cyberbullying Media-Based Prevention Intervention for Adolescents on Instagram: Pilot Randomized Controlled Trial. JMIR Ment Health. 2021 Sep 15;8(9):e26029. doi: 10.2196/26029. PMID 34524103